CLINICAL TRIAL: NCT02967094
Title: The Use of Mucolytic Solution Before Upper Endoscopy: A Randomized, Double-blinded Trial
Brief Title: Mucolytic Solution Before Upper Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vitkovice Hospital (Other)
Responsible Party: Principal Investigator, Premysl Falt, M.D., Ph.D., Principle Investigator, Vitkovice Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: DDC VN 09
Record Dates: First submitted 2016-11-10; First posted 2016-11-17 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Gastroscopy; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Espumisan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A - mucolytic solution (Experimental): Mucolytic solution consisting of 100 ml of water, 100 mg of simethicon and 400 mg of N-acetylcystein administered 30 minutes prior to upper endoscopy.
  Interventions: Drug: Administration of mucolytic solution before upper endoscopy (Espumisan, ACC long)
- B - no intervention (No Intervention): Upper endoscopy without neither mucolytic solution nor water prior to upper endoscopy.
- C - water (Placebo Comparator): 100 ml of water given 30 minutes prior to upper endoscopy.
  Interventions: Drug: Administration of water before upper endoscopy

INTERVENTIONS:
Drug: Administration of mucolytic solution before upper endoscopy (Espumisan, ACC long)
  Arms: A - mucolytic solution
Drug: Administration of water before upper endoscopy
  Arms: C - water

SUMMARY:
Study was designed to evaluate efficacy of mucolytic solution ingested before upper endoscopy on visibility of gastric mucosa.

DETAILED DESCRIPTION:
Residual gastric content containing mucus, bubbles, bile and food particles may limit visibility of gastric mucosa and therefore diagnostic yield of upper endoscopy, especially in cases of early neoplastic lesions. Data on benefit of peroral mucolytic solution administered before upper endoscopy are limited.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* signed informed consent
* diagnostic gastroscopy

Exclusion Criteria:

* age < 18 years
* interventional gastroscopy
* known disease of the upper GI tract and/or history of surgery of GI tract
* gastroscopy indicated of bleeding, dysphagia or ileus
* liver cirrhosis
* general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
"Visibility score" evaluated by blinded performing endoscopist | through study completion, an average of 3 months
  "Visibility score" (0-25 points) counted as the sum of visibility score in the esophagus (0-5), fundus (0-5), corpus (0-5) and atrum (0-5) of the stomach and in the duodenum (0-5).

SECONDARY OUTCOMES:
"Visibility score" evaluated by three blinded endoscopists using 11 endoscopic images captured during endoscopy. | through study completion, an average of 3 months
  "Visibility score" (0-25 points) counted as the sum of visibility score in the esophagus (0-5), fundus (0-5), corpus (0-5) and atrum (0-5) of the stomach and in the duodenum (0-5).
Residual fluid in the stomach evaluated by blinded performing endoscopist | through study completion, an average of 3 months
  0-3 point scale
Duration of endoscopy | through study completion, an average of 3 months
  time between introduction and withdrawal of the endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Premysl Falt, M.D., Ph.D., Principal Investigator — Digestive Diseases Center, Vítkovice Hospital
Locations (1):
- Digestive Diseases Center, Ostrava, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stepan M, Falt P, Pipek B, Fojtik P, Hanousek M, Hill M, Urban O. Administration of mucolytic solution before upper endoscopy - double-blind, monocentric, randomized study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2023 Mar;167(1):69-73. doi: 10.5507/bp.2021.038. Epub 2021 Jun 22. PMID 34158672